CLINICAL TRIAL: NCT00861614
Title: A Randomized, Double-Blind, Phase 3 Trial Comparing Ipilimumab vs. Placebo Following Radiotherapy in Subjects With Castration Resistant Prostate Cancer That Have Received Prior Treatment With Docetaxel
Brief Title: Study of Immunotherapy to Treat Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-043; 2008-003314-97
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab (Active Comparator)
  Interventions: Drug: Ipilimumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ipilimumab — 5 mg/ml solution, Intravenous, 10 mg/kg, Every 3 weeks for up to 4 doses in the Induction Phase. Every 12 weeks in the Maintenance Phase, Up to 24 weeks in Induction, 48+ weeks in the Maintenance Phase, or until Treatment Stopping Criteria are met, withdrawal of consent, lost to follow-up, death, study closure
  Other Names: BMS 734016
  Arms: Ipilimumab
Drug: Placebo — Solution, Intravenous, 0 mg, Every 3 weeks for up to 4 doses in the Induction Phase. Every 12 weeks in the Maintenance Phase, up to 24 weeks in Induction, 48+ weeks in the Maintenance Phase, or until Treatment Stopping Criteria are met, withdrawal of consent, lost to follow-up, death, study closure
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if advanced prostate cancer patients that are treated with radiotherapy (RT) plus ipilimumab live longer that those treated with RT alone

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Advanced prostate cancer
* At least 1 bone metastasis
* Testosterone < 50 ng/dl
* Prior treatment with docetaxel

Exclusion Criteria:

* Brain metastasis
* Autoimmune disease
* Known HIV, Hep B, or Hep C infection
* More than 2 prior systemic anticancer regimens for prostate cancer
* Prior treatment on BMS CA180227 for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 988 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (141):
- United States (44):
  - Southern Cancer Center, Mobile, Alabama
  - Alaska Clinical Research Center, Llc, Anchorage, Alaska
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Highlands Oncology Group, P.A., Fayetteville, Arkansas
  - Marsha G. Fink, Md, Inc., Fountain Valley, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - Prostate Oncology Specialists, Inc., Marina del Rey, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Va San Diego Healthcare System, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Baptist Cancer Institute, Jacksonville, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Suburban Hematology-Oncology Associates, Pc, Lawrenceville, Georgia
  - University Of Chicago, Chicago, Illinois
  - Cancer Care Specialists Of Central Illinois, Decatur, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Mid-Illinois Hematology & Oncology Associates, Ltd, Normal, Illinois
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Siouxland Hematology-Oncology Assoc., Llp, Sioux City, Iowa
  - Hutchinson Clinic, Pa, Hutchinson, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - The Bunting-Blaustein Cancer Research Building, Baltimore, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - St Johns Medical Research Institute, Inc., Springfield, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University Of Cincinnati, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - St. Luke'S Hospital & Health Network Laboratory, Bethlehem, Pennsylvania
  - Va Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Associates In Hematology & Oncology, P.C., Upland, Pennsylvania
  - Musc Hollings Cancer Center, Charleston, South Carolina
  - Center For Oncology Research & Treatment, P.A., Dallas, Texas
  - The Center For Cancer And Blood Disorders, Fort Worth, Texas
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
- Argentina (7):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Caba, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, La Rioja, La Rioja Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Australia (4):
  - Local Institution, Box Hill, Victoria
  - Local Institution, Frankston, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Subiaco, Western Australia
- Austria (2):
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Roeselare
- Brazil (8):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Curitiba, Paraná
  - Local Institution, Ijuí, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Curitiba, São Paulo
  - Local Institution, Divinopolis, São Paulo
  - Local Institution, Mogi das Cruzes, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (2):
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
- Chile (4):
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Vi?a Del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
  - Local Institution, Santiago - Independencia, Santiago Metropolitan
- Colombia (2):
  - Local Institution, Montería, Departamento de Córdoba
  - Local Institution, Bogotá
- Czechia (3):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Liberec
- Denmark (5):
  - Local Institution, Aalborg
  - Local Institution, Aarhus
  - Local Institution, Herlev
  - Local Institution, København Ø
  - Local Institution, Odense C
- France (6):
  - Local Institution, Besançon
  - Local Institution, Bordeaux
  - Local Institution, Clermont-Ferrand
  - Local Institution, Marseille
  - Local Institution, Pointe à Pitre
  - Local Institution, Villejuif
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Eschweiler
  - Local Institution, Mannheim
  - Local Institution, Wuppertal
- Local Institution, Athens, Greece
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Gyula
  - Local Institution, Kaposvár
  - Local Institution, Kecskemét
- Ireland (2):
  - Local Institution, Dublin, Dublin
  - Local Institution, Tallaght, Dublin
- Israel (5):
  - Local Institution, Beer Jacob
  - Local Institution, Beersheba
  - Local Institution, Haifa
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
- Italy (6):
  - Local Institution, Meldola (fc)
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Rimini
  - Local Institution, Siena
  - Local Institution, Sondrio
- Mexico (7):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Acapulco de Juárez, Guerrero
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Puebla City, Puebla
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Mb Amsterdam
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Arequipa
- Local Institution, Olsztyn, Poland
- Ponce School Of Medicine, Ponce, Puerto Rico
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Romania
  - Local Institution, Suceava
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Obninsk
  - Local Institution, Saint Petersburg
- Spain (5):
  - Local Institution, Barcelona
  - Local Institution, Benidorm-alicante
  - Local Institution, Madrid
  - Local Institution, Santiago de Compostela
  - Local Institution, Valencia
- United Kingdom (5):
  - Local Institution, Chelmsford, Essex
  - Local Institution, Cardiff, Glamorgan
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Scunthorpe, Lincolnshire
  - Local Institution, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Trump D. Commentary on: "Ipilimumab versus placebo after radiotherapy in patients with metastatic castration-resistant prostate cancer that had progressed after docetaxel chemotherapy (CA184-043): A multicentre, randomised, double-blind, phase 3 trial." Kwon ED, Drake CG, Scher HI, Fizazi K, Bossi A, van den Eertwegh AJ, Krainer M, Houede N, Santos R, Mahammedi H, Ng S, Maio M, Franke FA, Sundar S, Agarwal N, Bergman AM, Ciuleanu TE, Korbenfeld E, Sengelov L, Hansen S, Logothetis C, Beer TM, McHenry MB, Gagnier P, Liu D, Gerritsen WR, CA184-043 Investigators. Departments of Urology and Immunology and Mayo Clinic Comprehensive Cancer Center, Mayo Clinic, Rochester, MN, USA, Electronic address: kwon.eugene@mayo.edu; Johns Hopkins Sidney Kimmel Comprehensive Cancer Center and Brady Urological Institute, Baltimore, MD, USA; Memorial Sloan Kettering Cancer Center and Weill Cornell Medical College, New York, NY, USA; Institut Gustave Roussy, University of Paris-Sud, Villejuif, France; Institut Gustave Roussy, Villejuif, France; VU University Medical Centre, Amsterdam, Netherlands; Vienna General Hospital, Medical University Vienna, Vienna, Austria; Institut Bergonie, Bordeaux, France; CHU Caremeau, Nimes, France; Centro Medico Austral, Buenos Aires, Argentina; Centre Jean Perrin, Clermont-Ferrand, France; St John of God Hospital, Subiaco, WA, Australia; University Hospital of Siena, Istituto Toscano Tumori, Siena, Italy; Hospital de Caridade de Ijui, Ijui, Brazil; Nottingham University Hospital, Nottingham, UK; Huntsman Cancer Institute, University of Utah, Salt Lake City, UT, USA; Netherlands Cancer Institute and Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands; Institute of Oncology Ion Chiricuta and University of Medicine and Pharmacy Iuliu Hatieganu, Cluj-Napoca, Romania; Hospital Britanico de Buenos Aires, Buenos Aires, Argentina; Herlev Hospital, Herlev, Denmark; Odense University Hospital, Odense, Denmark; University of Texas MD Anderson Cancer Center, Houston, Urol Oncol. 2016 May;34(5):249-50. doi: 10.1016/j.urolonc.2015.03.013. Epub 2015 Apr 20. PMID 25907621
- [Derived] Kwon ED, Drake CG, Scher HI, Fizazi K, Bossi A, van den Eertwegh AJ, Krainer M, Houede N, Santos R, Mahammedi H, Ng S, Maio M, Franke FA, Sundar S, Agarwal N, Bergman AM, Ciuleanu TE, Korbenfeld E, Sengelov L, Hansen S, Logothetis C, Beer TM, McHenry MB, Gagnier P, Liu D, Gerritsen WR; CA184-043 Investigators. Ipilimumab versus placebo after radiotherapy in patients with metastatic castration-resistant prostate cancer that had progressed after docetaxel chemotherapy (CA184-043): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):700-12. doi: 10.1016/S1470-2045(14)70189-5. Epub 2014 May 13. PMID 24831977
- [Derived] Dayyani F, Gallick GE, Logothetis CJ, Corn PG. Novel therapies for metastatic castrate-resistant prostate cancer. J Natl Cancer Inst. 2011 Nov 16;103(22):1665-75. doi: 10.1093/jnci/djr362. Epub 2011 Sep 13. PMID 21917607
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 988 enrolled, 799 randomized (399 ipilimumab, 400 placebo); 149 no longer met study criteria, 17 withdrew, 6 adverse events, 4 died, 1 lost to follow-up,12 unspecified. 789 treated with radiotherapy (393 ipilimumab, 396 placebo); 2 no longer met study criteria, 3 withdrew consent, 1 died, 2 adverse events, 2 lost to follow-up.
Groups:
- Ipilimumab + Radiotherapy: Prior to receiving study drug, participants receive radiotherapy at 8 Gray units (Gy) to at least 1 and up to a maximum of 5, bone fields, all in one day. Within 2 days of radiotherapy, 10 milligrams (mg) of ipilimumab per kilogram (kg) of body weight was administered intravenously (IV) over 90 minutes. During the treatment phase, dosing was at weeks 1, 4, 7 and 10. In the maintenance phase, dosing was a 12-week intervals, beginning at week 24. Dosing continued until confirmed progressive disease (PD), drug intolerance, clinical deterioration, death, withdrawal of consent or subject lost to follow-up.
- Placebo + Radiotherapy: Prior to receiving study drug, participants receive radiotherapy at 8 Gy to at least 1 and up to a maximum of 5, bone fields, all in one day. Within 2 days of radiotherapy, placebo solution (0.9% sodium chloride or 5% dextrose) infused IV over 90 minutes. During the treatment phase, dosing was at weeks 1, 4, 7 and 10. In the maintenance phase, dosing was a 12-week intervals, beginning at week 24. Dosing continued until confirmed progressive disease (PD), drug intolerance, clinical deterioration, death, withdrawal of consent or subject lost to follow-up.
Period: Overall Study
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Started | 393 | 396
Completed | 22 | 28
Not Completed | 371 | 368
Not completed — Disease Progression | 182 | 263
Not completed — Study Drug Toxicity | 79 | 6
Not completed — Death | 32 | 19
Not completed — Adverse Event | 27 | 23
Not completed — Withdrawal by Subject | 34 | 35
Not completed — Other | 17 | 22

BASELINE CHARACTERISTICS:
Groups:
- Ipilimumab + Radiotherapy: Prior to receiving study drug, participants receive radiotherapy at 8 Gy to at least 1 and up to a maximum of 5, bone fields, all in one day. Within 2 days of radiotherapy, 10 milligrams (mg) of ipilimumab per kilogram (kg) of body weight was administered intravenously (IV) over 90 minutes. During the treatment phase, dosing was at weeks 1, 4,7 and 10. In the maintenance phase, dosing was a 12-week intervals, beginning at week 24. Dosing continued until confirmed progressive disease (PD), drug intolerance, clinical deterioration, death, withdrawal of consent or subject lost to follow-up.
- Placebo + Radiotherapy: Prior to receiving study drug, participants receive radiotherapy at 8 Gy to at least 1 and up to a maximum of 5, bone fields, all in one day. Within 2 days of radiotherapy, placebo solution (0.9% sodium chloride or 5% dextrose) infused IV over 90 minutes. During the treatment phase, dosing was at weeks 1, 4, 7 and 10. In the maintenance phase, dosing was a 12-week intervals, beginning at week 24. Dosing continued until confirmed PD, drug intolerance, clinical deterioration, death, withdrawal of consent or subject lost to follow-up.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy | Total
Number analyzed (Participants) | 399 | 400 | 799
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (7.53) | 67.1 (7.56) | 67.6 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 399 | 400 | 799

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time in months from randomization date to date of death due to any cause in all randomized subjects. For participants alive at the time of the database cutoff date, OS was censored at the last date the participant was known to be alive.
Time Frame: Date of randomization to date of death
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ipilimumab + Radiotherapy: Prior to receiving study drug, participants receive radiotherapy at 8 Gy to at least 1 and up to a maximum of 5, bone fields, all in one day. Within 2 days of radiotherapy, 10 milligrams (mg) of ipilimumab per kilogram (kg) of body weight was administered intravenously (IV) over 90 minutes. During the treatment phase, dosing was at weeks 1, 4, 7 and 10. In the maintenance phase, dosing was a 12-week intervals, beginning at week 24. Dosing continued until confirmed progressive disease (PD), drug intolerance, clinical deterioration, death, withdrawal of consent or subject lost to follow-up.
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 399 | 400
months | 11.04 [9.46 to 12.48] | 10.02 [8.38 to 11.17]
Statistical Analysis 1: Comparison: Ipilimumab + Radiotherapy vs Placebo + Radiotherapy; Test type: Superiority or Other; p = 0.0127, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.71 to 0.96] — Ipilimumab over placebo

2. Primary Outcome: Overall Survival Rate
Description: The overall survival (OS) rate is a percentage, representing the fraction of all randomized participants who were alive following treatment, from 1 to 5 years. OS was defined as the time between the date of randomization and the date of death as a result of any cause. Survival rates were determined via Kaplan-Meier estimates.
Time Frame: Date of randomization to date of death
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 399 | 400
percentage of participants
  OS Rate at Year 1 | 46.5 [41.6 to 51.4] | 40.8 [35.9 to 45.6]
  OS Rate at Year 2 | 25.2 [20.9 to 29.6] | 16.6 [12.9 to 20.3]
  OS Rate at Year 3 | 15.3 [11.7 to 18.9] | 7.9 [5.2 to 10.6]
  OS Rate at Year 4 | 10.1 [6.9 to 13.3] | 3.3 [1.3 to 5.3]
  OS Rate at Year 5 | 7.9 [4.4 to 11.4] | 2.7 [0.8 to 4.7]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: All PFS events were based on investigator's assessment. Participants who were alive and did not experience a PFS event were censored at the earlier of the latest prostate-specific antigen (PSA) or radiological tumor assessment date. Participants who did not die, showed no clinical deterioration, and who had no recorded post-baseline PSA or radiological tumor assessment were censored at randomization date.
Time Frame: Date of randomization to earliest date of confirmed PSA or radiological progression, clinical deterioration or death
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 399 | 400
months | 4.01 [3.65 to 4.34] | 3.06 [2.86 to 3.42]
Statistical Analysis 1: Comparison: Ipilimumab + Radiotherapy vs Placebo + Radiotherapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.61 to 0.82] — Ipilimumab over placebo

4. Secondary Outcome: Pain Response
Description: The percentage of participants with a pain response assessed using the Brief Pain Inventory Short Form (BPI-SF) completed by participants throughout the study in a daily diary log. Pain-evaluable participants were defined as those with a decrease in the average daily worst pain intensity by at least 30% from baseline, maintained over 2 consecutive evaluations without the use of any rescue analgesic medication or increase in analgesic use in the same time period.
Time Frame: Assessed at screening, weeks 12, 18, 24, and at the end of treatment visit
Population: All pain-evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 197 | 186
percentage of participants | 3.55 [1.44 to 7.18] | 0.54 [0.01 to 2.96]

5. Secondary Outcome: Duration of Pain Response
Description: The time between the initial date of pain response and completion date of pain response. The initial date when the pain response criterion was achieved was considered the pain response date. The earlier of date of death, date of tumor resection surgery, or date when pain response criterion was no longer met was considered the completion date of the pain response. If none of these scenarios occurred, the completion of the pain response was set to the last known alive date.
Time Frame: Day of initial pain response to day of completion of pain response or date of death
Population: All pain-evaluable participants with pain response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 7 | 1
months | 2.5 [1.5 to 3] | 1.5 [NA to NA] — CI not applicable due to only one participant
Statistical Analysis 1: Comparison: Ipilimumab + Radiotherapy vs Placebo + Radiotherapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.02 to 4.00] — Ipilimumab over placebo

6. Secondary Outcome: Number of Participants With Severe Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths, Discontinuation of Study Drug Due to AEs, Immune-Related Adverse Events (irAE) and Immune-Mediated Adverse Reaction (imAR)
Description: AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment.
  SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during study and up to 70 days after last dose. IrAEs=AEs potentially associated with inflammation and considered to be causally related to study drug and grouped into gastrointestinal (GI), hepatic, skin, endocrine and neurological. ImARs were collected prospectively and grouped into enterocolitis, hepatitis, dermatitis, neuropathies and endocrinopathies. IrAEs/ imARs were graded using Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), Ver. 3.0.
Time Frame: Randomization to date of death
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
participants
  SAE | 257 | 164
  Treatment-Related AE | 296 | 180
  Any Death | 346 | 371
  Deaths Due to Study Drug Toxicity | 7 | 1
  Discontinuation of Study Drug due to AEs | 137 | 62
  Immune-Related AE (any grade) | 250 | 86
  Immune-Mediated Adverse Reaction (Grade >=2) | 203 | 40

7. Secondary Outcome: Time to Onset of Grade 3 or 4 Immune-Related Adverse Event (irAE)
Description: The time between first dose of study drug and date of earliest Grade 3 or 4 irAE. These irAEs are AEs of unknown etiology, consistent with an immune phenomenon and considered as causally related to drug exposure. The five subcategories of irAE examined include gastrointestinal (GI), liver, skin, endocrine, and neurological and are graded using the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
weeks
  Gastrotintestinal (n= 71,3) | 5.71 [5.00 to 7.00] | 5.71 [0.57 to 31.86]
  Liver (n= 18,5) | 9.14 [8.29 to 10.43] | 6.00 [3.14 to 8.57]
  Skin (n=4,0) | 3.71 [2.57 to 6.43] | NA [NA to NA] — There were no participants in this treatment arm who displayed irAEs of this type
  Endocrine (n=8,2) | 7.93 [4.14 to 11.14] | 5.00 [4.29 to 5.71]
  Neurological (n= 1,0) | 11.4 [NA to NA] — CI not applicable due to only one participant | NA [NA to NA] — There were no participants in this treatment arm who displayed irAEs of this type

8. Secondary Outcome: Time to Resolution of Grade 3 or 4 Immune-Related Adverse Event (irAE)
Description: Time between the date of onset of a Grade 3 or 4 irAE and the date of improvement to Grade 1 or less or the worst grade at baseline.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
weeks
  Gastrointestinal (n=71,3) | 2.9 [1.6 to 4.7] | 0.9 [0.4 to 1.1]
  Liver (n=18,5) | 4.1 [3.6 to 8.1] | 6.0 [1.9 to NA] — Number of subjects was too small to obtain upper limit
  Skin (n=4,0) | 3.6 [2.6 to 5.9] | NA [NA to NA] — There were no participants in this treatment arm who displayed irAEs of this type.
  Endocrine (n=8,2) | 11.1 [2.4 to NA] — Number of subjects was too small to obtain upper limit | 5.9 [0.9 to 10.9]
  Neurological (n=1,0) | NA [NA to NA] — No participant with resolved irAE. | NA [NA to NA] — There were no participants in this treatment arm who displayed irAEs of this type.

9. Secondary Outcome: Time to Onset of Grade 3 to 5 Immune-Mediated Adverse Reaction (imAR)
Description: The time between first dose of study drug and date of earliest Grade 3 or 4 imAR. ImARs were collected prospectively and grouped into enterocolitis, hepatitis, dermatitis, neuropathies and endocrinopathies and graded using Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), Ver. 3.0.
  Only the Ipilimumab + Radiotherapy group of participants was included in the analysis because ipilimumab is associated with inflammatory events resulting from increased or excessive immune activity likely to be related to its mechanism of action.
Time Frame: Day 1 to time of onset of the imAR of interest
Population: All treated participants receiving Ipilimumab + Radiotherapy
Measure: Median (Full Range); unit: weeks
Arm/Group | Ipilimumab + Radiotherapy
Number analyzed (Participants) | 393
weeks
  Enterocolitis (n=65) | 3.4 [0.3 to 16.6]
  Hepatitis (n=17) | 9.0 [1.7 to 16.9]
  Dermatitis (n=3) | 2.4 [0.1 to 3.1]
  Endocrinopathies (n=6) | 7.9 [1.7 to 10.7]

10. Secondary Outcome: Time to Resolution of Grade 3 to 5 to Grade 0 Immune-Mediated Adverse Reactions (imARs) to Grade 0
Description: Time between the date of onset of an imAR to the date of resolution date of the event or the last known date participant was alive if an event did not resolve.
  Only the Ipilimumab + Radiotherapy group of participants was included in the analysis because ipilimumab is associated with inflammatory events resulting from increased or excessive immune activity likely to be related to its mechanism of action.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants receiving Ipilimumab + Radiotherapy
Measure: Median (Full Range); unit: weeks
Arm/Group | Ipilimumab + Radiotherapy
Number analyzed (Participants) | 393
weeks
  Enterocolitis (n=52) | 6.0 [0.1 to 40.1]
  Hepatitis (n=15) | 8.6 [1.1 to 19.0]
  Dermatitis (n=3) | 6.9 [4.0 to 12.1]
  Endocrinopathies (n=0) | NA [NA to NA] — No participant with resolved imAR

11. Secondary Outcome: Number of Participants With Worst On-Study Hematology Common Toxicity Criteria (CTC) Grade and Shift From Baseline
Description: Comparison of baseline versus worst grade hematology laboratory tests as measured by white blood count (WBC), absolute neutrophil count (ANC), platelet count, hemoglobin and lymphocyte results. National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade (Gr). Gr 0: within normal range. Abnormal values for WBC were based on Gr 1: 3.0 - < Lower Limit of Normal (LLN); Gr 2: 2.0 - < 3.0; Gr 3: 1.0 - < 2.0; Gr4: < 1.0. Abnormal values for Hemoglobin were based on Gr 1: 10.0 - < LLN; Gr 2: 8.0 - < 10.0; Gr 3: 6.5 - < 8.0; Gr 4: < 6.5. Abnormal values for Lymphocytes were based on Gr 1: 0.8 - < 1.5; Gr 2: 0.5 - < 0.8; Gr 3): 0.2 - < 0.5; Gr 4: < 0.2. Abnormal values for ANC were based on Gr 1: 1.5 - < 2.0; Gr 2: 1.0 - < 1.5; Gr 3: 0.5 - < 1.0; Gr 4: < 0.5. Abnormal values for Platelets were based on Gr 1: 75.0 - < LLN; Gr 2: 50.0 - < 75.0; Gr 3: 25.0 - < 50.0; Gr 4: < 25.0.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
participants
  WBC Gr 0 at Baseline to Gr 3-4 | 3 | 2
  WBC Gr 1 at Baseline to Gr 3-4 | 0 | 1
  WBC Gr 2 at Baseline to Gr 3-4 | 0 | 1
  WBC Gr 3 at Baseline to Gr 3-4 | 0 | 0
  WBC Gr 4 at Baseline to Gr 3-4 | 0 | 0
  WBC Not Reported at Baseline to Gr 3-4 | 0 | 0
  ANC Gr 0 at Baseline to Gr 3-4 | 4 | 6
  ANC Gr 1 at Baseline to Gr 3-4 | 0 | 0
  ANC Gr 2 at Baseline to Gr 3-4 | 0 | 0
  ANC Gr 3 at Baseline to Gr 3-4 | 0 | 0
  ANC Gr 4 at Baseline to Gr 3-4 | 0 | 0
  ANC Not Reported at Baseline to Gr 3-4 | 1 | 0
  Platelet Count Gr 0 at Baseline to Gr 3-4 | 1 | 6
  Platelet Count Gr 1 at Baseline to Gr 3-4 | 1 | 1
  Platelet Count Gr 2 at Baseline to Gr 3-4 | 0 | 0
  Platelet Count Gr 3 at Baseline to Gr 3-4 | 0 | 0
  Platelet Count Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Platelet Count Not Reported at Baseline to Gr 3-4 | 1 | 1
  Hemoglobin Gr 0 at Baseline to Gr 3-4 | 0 | 3
  Hemoglobin Gr 1 at Baseline to Gr 3-4 | 16 | 25
  Hemoglobin Gr 2 at Baseline to Gr 3-4 | 13 | 11
  Hemoglobin Gr 3 at Baseline to Gr 3-4 | 0 | 1
  Hemoglobin Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Hemoglobin Not Reported at Baseline to Gr 3-4 | 0 | 1
  Lymphocytes Gr 0 at Baseline to Gr 3-4 | 4 | 1
  Lymphocytes Gr 1 at Baseline to Gr 3-4 | 6 | 11
  Lymphocytes Gr 2 at Baseline to Gr 3-4 | 11 | 17
  Lymphocytes Gr 3 at Baseline to Gr 3-4 | 8 | 7
  Lymphocytes Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Lymphocytes Not Reported at Baseline to Gr 3-4 | 3 | 0

12. Secondary Outcome: Number of Participants With Worst On-Study Liver Common Toxicity Criteria (CTC) Grade and Shift From Baseline
Description: Comparison of baseline versus worst grade liver function as measured by alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin and alkaline phosphatase (ALP). National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade (Gr). Gr 0: within normal range. Abnormal values for ALP, ALT and AST were based on grades; Gr 1: > 1.0 - 2.5 * upper limits of normal (ULN); Gr 2: > 2.5 - 5.0 * ULN; Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Abnormal values for Total Bilirubin were based on Gr 1: > 1.0 - 1.5 * upper limits of normal (ULN); Gr 2: > 1.5 - 3.0 * ULN; Gr 3: > 3.0 - 10.0 * ULN; Gr 4: > 10.0 * ULN.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
participants
  ALT Gr 0 at Baseline to Gr 3-4 | 16 | 1
  ALT Gr 1 at Baseline to Gr 3-4 | 1 | 1
  ALT Gr 2 at Baseline to Gr 3-4 | 0 | 0
  ALT Gr 3 at Baseline to Gr 3-4 | 0 | 0
  ALT Gr 4 at Baseline to Gr 3-4 | 0 | 0
  ALT Not reported at Basline to Gr 3-4 | 1 | 0
  AST Gr 0 at Baseline to Gr 3-4 | 15 | 6
  AST Gr 1 at Baseline to Gr 3-4 | 5 | 1
  AST Gr 2 at Baseline to Gr 3-4 | 1 | 1
  AST Gr 3 at Baseline to Gr 3-4 | 1 | 0
  AST Gr 4 at Baseline to Gr 3-4 | 0 | 0
  AST Not Reported at Baseline to Gr 3-4 | 1 | 0
  Total Bilirubin Gr 0 at Baseline to Gr 3-4 | 6 | 2
  Total Bilirubin Gr 1 at Baseline to Gr 3-4 | 1 | 0
  Total Bilirubin Gr 2 at Baseline to Gr 3-4 | 1 | 0
  Total Bilirubin Gr 3 at Baseline to Gr 3-4 | 0 | 0
  Total Bilirubin Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Total Bilirubin Not Reported at Baseline to Gr 3-4 | 0 | 0
  ALP Gr 0 at Baseline to Gr 3-4 | 1 | 1
  ALP Gr 1 at Baseline to Gr 3-4 | 10 | 17
  ALP Gr 2 at Baseline to Gr 3-4 | 21 | 29
  ALP Gr 3 at Baseline to Gr 3-4 | 27 | 42
  ALP Gr 4 at Baseline to Gr 3-4 | 1 | 0
  ALP Not Reported at Baseline to Gr 3-4 | 0 | 6

13. Secondary Outcome: Number of Participants With Worst On-Study Serum Chemistry Common Toxicity Criteria (CTC) Grade and Shift From Baseline
Description: Comparison of baseline versus worst grade serum chemistry as measured by lipase and amylase analysis. National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade (Gr). Gr 0: within normal range. Abnormal values for lipase: Gr1: > 1.0 - 1.5 * ULN; Gr2: > 1.5 - 2.0 * ULN; Gr 3: > 2.0 - 5.0 * ULN; Gr4: > 5.0*ULN. Abnormal values for amylase: Gr1: > 1.0 - 1.5 * ULN; Gr 2: > 1.5 - 2.0 * ULN; Gr 3: > 2.0 - 5.0 * ULN; Gr4: > 5.0 * ULN.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
participants
  Lipase Gr 0 at Baseline to Gr 3-4 | 21 | 10
  Lipase Gr 1 at Baseline to Gr 3-4 | 1 | 1
  Lipase Gr 2 at Baseline to Gr 3-4 | 1 | 0
  Lipase Gr 3 at Baseline to Gr 3-4 | 0 | 1
  Lipase Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Lipase Not reported at Basline to Gr 3-4 | 0 | 0
  Amylase Gr 0 at Baseline to Gr 3-4 | 4 | 4
  Amylase Gr 1 at Baseline to Gr 3-4 | 1 | 1
  Amylase Gr 2 at Baseline to Gr 3-4 | 3 | 1
  Amylase Gr 3 at Baseline to Gr 3-4 | 1 | 0
  Amylase Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Amylase Not Reported at Baseline to Gr 3-4 | 0 | 0

14. Secondary Outcome: Number of Participants With Worst On-Study Renal Function Common Toxicity Criteria (CTC) Grade and Shift From Baseline
Description: Comparison of baseline versus worst grade renal function as measured by creatinine analysis. National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade (Gr).Gr 0: within normal range. Abnormal values for Creatinine were based on Gr 1: > 1.0 - 1.5*ULN; Gr 2: > 1.5 - 3.0*ULN; Gr 3: > 3.0 - 6.0*ULN; Gr 4: > 6.0*ULN.
Time Frame: Day 1 to 70 days after last dose of study drug
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Number analyzed (Participants) | 393 | 396
participants
  Creatinine Gr 0 at Baseline to Gr 3-4 | 3 | 3
  Creatinine Gr 1 at Baseline to Gr 3-4 | 0 | 0
  Creatinine Gr 2 at Baseline to Gr 3-4 | 0 | 0
  Creatinine Gr 3 at Baseline to Gr 3-4 | 0 | 0
  Creatinine Gr 4 at Baseline to Gr 3-4 | 0 | 0
  Creatinine Not Reported at Baseline to Gr 3-4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to 70 days following the last dose of study drug
Description: Study initiated: May 2009; Study completed: August 2015
Arm/Group | Ipilimumab + Radiotherapy | Placebo + Radiotherapy
Serious Adverse Events (participants affected / at risk) | 257/393 | 164/396
Other Adverse Events (participants affected / at risk) | 350/393 | 333/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + Radiotherapy (N=393) | Placebo + Radiotherapy (N=396)
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 18 | 10
Depression (Psychiatric disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
General physical health deterioration (General disorders) | 16 | 8
Hallucination (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Hepatitis (Hepatobiliary disorders) | 4 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 4 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Self injurious behaviour (Psychiatric disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2
Central nervous system infection (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 21 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypophysitis (Endocrine disorders) | 2 | 2
Hypothyroidism (Endocrine disorders) | 2 | 0
Lethargy (Nervous system disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Malaise (General disorders) | 7 | 1
Mucosal inflammation (General disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Pneumonia (Infections and infestations) | 18 | 5
Renal impairment (Renal and urinary disorders) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bladder dilatation (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1
C-reactive protein increased (Investigations) | 1 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 2
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 2
Confusional state (Psychiatric disorders) | 3 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Fatigue (General disorders) | 13 | 10
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Liver function test abnormal (Investigations) | 3 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Paresis (Nervous system disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pupils unequal (Eye disorders) | 0 | 1
Pyrexia (General disorders) | 17 | 2
Red blood cell count decreased (Investigations) | 0 | 1
Renal injury (Renal and urinary disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cavernous sinus thrombosis (Infections and infestations) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 2
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 13 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hypopituitarism (Endocrine disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nausea (Gastrointestinal disorders) | 11 | 8
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Papilloedema (Eye disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Anal infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Blood creatine phosphokinase decreased (Investigations) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 59 | 6
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Spinal cord compression (Nervous system disorders) | 4 | 2
Spinal cord infection (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 2
Venous thrombosis (Vascular disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2
Bronchopneumonia (Infections and infestations) | 0 | 3
Cardiac valve disease (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 2 | 3
Chills (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 | 31
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6
Thrombosis (Vascular disorders) | 1 | 0
Tongue paralysis (Nervous system disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Urinary tract infection (Infections and infestations) | 12 | 4
Vomiting (Gastrointestinal disorders) | 11 | 10
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 2
Anaemia (Blood and lymphatic system disorders) | 15 | 18
Asthenia (General disorders) | 9 | 4
Autoimmune disorder (Immune system disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Haematuria (Renal and urinary disorders) | 6 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain (General disorders) | 6 | 10
Performance status decreased (General disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Syncope (Nervous system disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 2 | 2
Urosepsis (Infections and infestations) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 0
Arrhythmia (Cardiac disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Brachial plexopathy (Nervous system disorders) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
General physical condition abnormal (Investigations) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 1
Infection (Infections and infestations) | 2 | 2
Macular degeneration (Eye disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 0
Multi-organ failure (General disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 6 | 3
Somnolence (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Weight decreased (Investigations) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + Radiotherapy (N=393) | Placebo + Radiotherapy (N=396)
Dehydration (Metabolism and nutrition disorders) | 26 | 15
Depression (Psychiatric disorders) | 10 | 20
Headache (Nervous system disorders) | 38 | 31
Abdominal pain (Gastrointestinal disorders) | 33 | 25
Decreased appetite (Metabolism and nutrition disorders) | 119 | 97
Hypertension (Vascular disorders) | 20 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 10
Insomnia (Psychiatric disorders) | 31 | 34
Pruritus (Skin and subcutaneous tissue disorders) | 99 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 27
Dizziness (Nervous system disorders) | 22 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 32
Fatigue (General disorders) | 144 | 120
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32 | 44
Oedema peripheral (General disorders) | 46 | 33
Pyrexia (General disorders) | 81 | 50
Aspartate aminotransferase increased (Investigations) | 31 | 21
Haemoglobin decreased (Investigations) | 26 | 20
Nausea (Gastrointestinal disorders) | 126 | 104
Rash (Skin and subcutaneous tissue disorders) | 81 | 27
Diarrhoea (Gastrointestinal disorders) | 186 | 94
Constipation (Gastrointestinal disorders) | 66 | 82
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 41
Urinary tract infection (Infections and infestations) | 24 | 24
Vomiting (Gastrointestinal disorders) | 107 | 80
Anaemia (Blood and lymphatic system disorders) | 79 | 81
Asthenia (General disorders) | 80 | 64
Pain (General disorders) | 33 | 44
Alanine aminotransferase increased (Investigations) | 26 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 57
Back pain (Musculoskeletal and connective tissue disorders) | 56 | 74
Bone pain (Musculoskeletal and connective tissue disorders) | 31 | 53
Weight decreased (Investigations) | 91 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less